CLINICAL TRIAL: NCT01487980
Title: The Effect of Delayed Cord Clamping on Haematological Status in Low Birth Weight Infants: a Randomised Controlled Trial in South Africa.
Brief Title: Effect of Delayed Cord Clamping on Haematological Status in Low Birth Weight Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanger Hospital (Other)
Collaborators: Otto Kranendonk Fonds - Dutch Association of Tropical Health (request pending) (Unknown)
Responsible Party: Principal Investigator, S. Tiemersma, Medical Officer, Stanger Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: DCC-LBW-SA
Record Dates: First submitted 2011-12-05; First posted 2011-12-08 (Estimated); Last update posted 2012-12-18 (Estimated); Status verified 2012-12

CONDITIONS: Low Birth Weight; Perinatology; Iron Status; Cord Clamping
MeSH Terms: interventions — Umbilical Cord Clamping

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early cord clamping (Active Comparator): Within 30 seconds after birth.
  Interventions: Procedure: Cord clamping
- Delayed cord clamping (Experimental): Between 2 and 3 minutes after birth
  Interventions: Procedure: Cord clamping

INTERVENTIONS:
Procedure: Cord clamping — Early vs Delayed

SUMMARY:
Delayed cord clamping (DCC, clamping after cessation of pulsations in the cord around 2-3 min after delivery) is effective in increasing (low birth weight) infant haemoglobin and iron status until six months after birth, without increasing the risk of polycythaemia or other adverse events. We hypothesize that this intervention will also benefit low birth weight infants in South Africa.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant mothers with SFH measurements below the cutpoint are eligible for inclusion. We aim to include infants with a birth weight below 2500 grams, but the actual birthweight can only be assessed after birth. We therefore accept an error of 500 grams (20%) and will include newborns up to 3000 grams. Birthweight will be measured after randomisation and study treatment.

Exclusion Criteria:

1. twin pregnancy
2. history of postpartum haemorrhage (PPH)
3. (gestational) diabetes
4. pre-eclampsia
5. abruptio placentae
6. caesarian section
7. necessity of early clamping due to tight nuchal cord
8. need for resuscitation immediately after birth
9. major congenital abnormalities

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Estimated)
Dates: Start 2012-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Haemoglobin level | two months

SECONDARY OUTCOMES:
Hyperviscosity syndrome | 1 day
Iron status | two months
hyperbilirubinaemia | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Sybrich Tiemersma, MD, Principal Investigator — Stanger Hospital
Locations (1):
- Stanger Hospital, KwaDukuza, KwaZulu-Natal, South Africa